CLINICAL TRIAL: NCT01114815
Title: Natural History of CADASIL: Migraine, Diagnosis and Misdiagnosis
Brief Title: Research Study on Cerebral Autosomal Dominant Arteriopathy With Subcortical Infarcts and Leukoencephalopathy (CADASIL)
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: NYU IRB #09-0214
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: CADASIL
Keywords: CADASIL; cerebral; autosomal dominant; arteriopathy; subcortical infarcts; leukoencephalopathy
MeSH Terms: conditions — CADASIL; Multiple Pterygium Syndrome, Autosomal Dominant; Leukoencephalopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to delineate early neurological features and their progression in patients with cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL) in order to facilitate early diagnosis, prevent erroneous diagnosis and mistreatment and improve physician education about this relatively common yet under-recognized dementing disorder.

Patients with CADASIL suffer from a variant from migraine that differs from wild type migraine in terms of its severity, progressive nature and underlying pathophysiology. Recurrent stereotypic acute confusional state associated with the headache episodes in patients with CADASIL is a distinctive phenomenon, which if recognized will lead to an earlier and accurate diagnosis of this condition.

Specific Aims:

* Characterize the nature, frequency and severity of migraine in patients with CADASIL.
* Delineate the phenomenon of acute confusional migraine as a distinct subgroup of migraine and establish its prevalence in patients with CADASIL.
* Determine the latency between the onset of neurological symptoms including migraine, and diagnosis of CADASIL and the prevalence of misdiagnosis.

DETAILED DESCRIPTION:
New York University School of Medicine, Division of Neurogenetics is conducting a new research study for patients with CADASIL (cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy). We are inviting anyone age 18 or older with a confirmed diagnosis of CADASIL to participate. We greatly appreciate your help in this regard. Please be assured that if you participate, all the information you, your relatives or your physicians provide will be held in strict confidence.

CADASIL is often misdiagnosed due to lack of awareness of this condition among health care providers and because the disease can closely mimic other neurological conditions. People with CADASIL struggle to find a doctor who has knowledge about this condition. The purpose of this study is to better understand the early symptoms of CADASIL so doctors may learn to diagnose it early.

This research study will be based on review of medical information provided by you or your health care giver. If you are interested, please contact us by telephone. We will mail a questionnaire for you to fill out and return to us, and request a copy of your brain MRI, test results and office notes from your doctor. We will contact some people for a more detailed telephone interview. Your responses and questionnaire are still valuable even if we do not get other records. The estimated time to complete the questionnaire is about two hours. The telephone interview (if applicable) is expected to last for 30 to 45 minutes. It may be helpful to involve a family member or a friend while completing the questionnaire.

If you wish to participate in this study, please call our research office.We will tell you about the project and then, if you wish to participate, will mail you the questionnaires with return envelopes. Your participation and support is deeply appreciated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CADASIL confirmed by Notch3 sequencing and/or skin biopsy.
* Age: 18+
* Subjects with speech, motor and/ or cognitive impairment will be included if their surrogate can provide the necessary information.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone with confirmed diagnosis of CADASIL
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To distinguish between CADASIL subjects with migraine and without migraine | Retrospective data was collected- cross sectional case control study- history of migraine until the time of enrollment was collected
  We sent a questionnaire to CADASIL subjects upon their consent to enroll in the study. The questionnaire addressed the history of migraine in till the time of enrollment. Other features such as history of stroke, memory involvement till enrollment was assessed in the questionnaire. The study aims at comparing the two groups- subjects with migraine and without migraine.

CONTACTS AND LOCATIONS:
Overall Officials: Swati A Sathe, MD, MS, Principal Investigator — NYU School of Medicine, Division of Neurogenetics
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Chabriat H, Vahedi K, Iba-Zizen MT, Joutel A, Nibbio A, Nagy TG, Krebs MO, Julien J, Dubois B, Ducrocq X, et al. Clinical spectrum of CADASIL: a study of 7 families. Cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy. Lancet. 1995 Oct 7;346(8980):934-9. doi: 10.1016/s0140-6736(95)91557-5. PMID 7564728
- [Background] Desmond DW, Moroney JT, Lynch T, Chan S, Chin SS, Mohr JP. The natural history of CADASIL: a pooled analysis of previously published cases. Stroke. 1999 Jun;30(6):1230-3. doi: 10.1161/01.str.30.6.1230. PMID 10356105
- [Background] Vahedi K, Chabriat H, Levy C, Joutel A, Tournier-Lasserve E, Bousser MG. Migraine with aura and brain magnetic resonance imaging abnormalities in patients with CADASIL. Arch Neurol. 2004 Aug;61(8):1237-40. doi: 10.1001/archneur.61.8.1237. PMID 15313840
- [Background] Sathe S, DePeralta E, Pastores G, Kolodny EH. Acute confusional migraine may be a presenting feature of CADASIL. Headache. 2009 Apr;49(4):590-6. doi: 10.1111/j.1526-4610.2009.01363.x. Epub 2009 Feb 25. PMID 19245392